CLINICAL TRIAL: NCT05907967
Title: A Randomized, Double Blind Sham Controlled Clinical Trial to Evaluate The Efficacy of Electrical Vestibular Stimulation (VeNS), Compared to a Sham Control For The Management Of Anxiety
Brief Title: Electrical Vestibular Stimulation (VeNS), Compared to a Sham Control For The Management Of Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovalens Ltd. (Industry)
Collaborators: Ulster University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UUS002
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active VeNS (Active Comparator): The active device utilizes a technology termed vestibular nerve stimulation (VeNS). The device will be placed on the head in a manner analogous to headphones and will deliver a small electrical current to the skin behind the ears, over the mastoid processes. Participants will be advised to use the device at home for 30 minutes per day.
  Interventions: Device: VeNS
- Sham VeNS (Sham Comparator): The sham device looks identical to the active device and interacts with the app in a similar manner to the active device. It will apply some stimulation to a user for a limited period of time (30 seconds), before tapering down to zero over a further 20 seconds, thus creating the impression of an active device. The device will be placed on the head in a manner analogous to headphones with hydrogel electrodes placed over the mastoid processes. Participants will be advised to use the device at home for 30 minutes per day.
  Interventions: Device: VeNS

INTERVENTIONS:
Device: VeNS — The VeNS device utilizes a technology called galvanic vestibular stimulation (GVS) (sometimes termed vestibular nerve stimulation (VeNS)). The device will be placed on the head in a manner analogous to headphones and will deliver a small electrical current to the skin behind the ears, over the mastoid processes. Participants will be advised to use the device at home for 30 minutes per day.

SUMMARY:
Anxiety is known to be one of the most common health concerns in in the general population, and the most common mental health issue, and has been associated with several health consequences. Medications are known to be effective, and currently serve as the primary treatment for anxiety but comes with a risk of adverse effects. Cognitive Behavioral Therapy (CBT-1) has also been shown to be effective and safer in the treatment of anxiety but presents its own limitations such as the time, cost, and training required. The relationship between vestibular stimulation and anxiety continues to be explored, however its usefulness in the treatment of anxiety is still unknown. Vestibular stimulation itself has been shown to be safe across multiple populations. If vestibular stimulation is shown to be effective in the treatment of anxiety, it could serve as a safer alternative to medications. It could also require less cost, time, and training than CBT-1, providing a treatment option that is not only safe and effective, but broadly available to the general population. It also could present an alternative intervention for patients who are non-responsive or refuse medication. Consequently this trial seeks to evaluate the efficacy of non-invasive electrical vestibular nerve stimulation as a method of improving sleep quality and quantity, as compared to a sham control, in patients newly diagnosed with anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male or female, age ≥ 18 years and ≤ 80 years at the time of signing informed consent.
* Report clinically significant symptoms of anxiety, defined as a score of 10 or greater on the Generalized Anxiety Disorder Scale, 7th edition (GAD-7)
* Ability and willingness to complete all study visits and procedures
* Agreement to engage with using the device on a daily basis
* Agreement to engage with trial mentors
* Agreement not to use prescription, or over the counter, anxiety medications for the duration of the trial
* Access to Wi-Fi
* Access to Apple smart phone (If not an Apple iPod will be supplied)

Exclusion Criteria:

* History of skin breakdown, eczema or other dermatological condition (e.g. psoriasis) affecting the skin behind the ears.
* Previous diagnosis of HIV infection or AIDS (HIV is known to cause a vestibular neuropathy which would prevent VeNS from working)
* Use of beta-blockers within 1 month of starting the study
* Use of antidepressants or unstable dose within 3 months of starting study
* Medication for anxiety (unless regime stable for last 3 months).
* A history of stroke or severe head injury (as defined by a head injury that required a craniotomy or endotracheal intubation). (In case this damaged the neurological pathways involved in vestibular stimulation).
* Presence of permanently implanted battery powered medical device or stimulator (e.g., pacemaker, implanted defibrillator, deep brain stimulator, vagal nerve stimulator etc.).
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice)
* History of epilepsy
* History of active migraines with aura
* History of head injury requiring intensive care or neurosurgery
* History of cognitive impairment
* History of of bipolar, psychotic or substance use disorders
* Regular use (more than twice a month) of antihistamine medication within the last 6 months.
* History or presence of malignancy within the last year (except basal and squamous cell skin cancer and in-situ carcinomas)
* A diagnosis of myelofibrosis or a myelodysplastic syndrome.
* Previous use of Modius device
* Participation in other clinical trials sponsored by Neurovalens
* Participation in any other anxiety studies
* Have a member of the same household who is currently participating in this study.
* Not fluent in English language
* History of vestibular dysfunction or other inner ear disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Generalised Anxiety Disorder (GAD-7) Scores | 4 weeks
  To evaluate the effect of the VeNS device, relative to control group on participants with anxiety (range 0-21) with higher score indicating more severe anxiety.

SECONDARY OUTCOMES:
Number of adverse events | 4 weeks
  To evaluate the safety of the VeNS device relative to control group, in terms of the occurrence of adverse events.
Quality of life using SF-36 scores | 4 weeks
  To evaluate the effect of the VeNS device, relative to control group, on quality of life. SF-36 is a 36-item short form survey (range 0-100) with higher scores indicating a better quality of life.
Insomnia Severity Index (ISI) score | 4 weeks
  To evaluate the effect of the VeNS device, relative to control group on participants with insomnia. ISI is a self-report rating scale assessing the severity of insomnia symptoms (range 0-28) with higher scores indicating a more severe insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Sittlington, PhD, Principal Investigator — Ulster University
Locations (1):
- Ulster University, Coleraine, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Curry G, Zhang SD, McAnena L, Price RK, Sittlington JJ. Repeated Electrical Vestibular Nerve Stimulation Reduces Anxiety in People With Moderate-to-Severe Anxiety: A Randomized, Sham-Controlled Trial: The Modius Anxiety Study. Neuromodulation. 2026 Feb 5:S1094-7159(25)01152-3. doi: 10.1016/j.neurom.2025.11.008. Online ahead of print. PMID 41642155